CLINICAL TRIAL: NCT00175968
Title: Influence of Bed-Rest and Hypocaloric Nutrition on Endothelium-Dependent Vasoreactivity
Brief Title: Influence of Bedrest and Hypocaloric Nutrition on Endothelium-Dependent Vasoreactivity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Heidelberg University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Educational/Counseling/Training
Other Study IDs: K008
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-09

CONDITIONS: Healthy
MeSH Terms: interventions — Bed Rest

INTERVENTIONS:
Procedure: bed rest, hypocaloric nutrition

SUMMARY:
Aim of the study is to assess the impact of the factors ´bed rest´ and ´hypocaloric nutrition´ on endothelium-dependent vasoreactivity in healthy volunteers.

DETAILED DESCRIPTION:
In a randomized, four-phase cross-over study the effect of simulated microgravity (13 days of bed rest), energetic restriction (-25%, fat reduced), and their combination on endothelium-dependent and -independent vasodilation will be compared with ambulatory control conditions. Using venous occlusion plethysmography cumulative intraarterial dose-response curves to endothelium-dependent (acetylcholine) and -independent (sodium nitroprusside) vasodilators will be constructed in 10 healthy male volunteers before and on day 13 of each of the four intervention periods.

ELIGIBILITY:
Inclusion Criteria:´

* Healthy, male volunteers, age: 18-40
* Able and willing to give written informed consent

Exclusion Criteria:

* Known condition causing endothelial dysfunction (e.g. diabetes, hyperlipidaemia, arterial hypertension, smoking, hyperhomocysteinaemia)
* Regular medication and/or treatment with drugs within the last 4-6 weeks (exclusion has to be decided in each case)
* Acute or chronic illness
* Participation in clinical trial/blood donation within 2 month before the study
* Nicotine during 1 year before the study; drug and/or alcohol abuse.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10
Dates: Start 2001-03; Study Completion 2003-04

PRIMARY OUTCOMES:
Drug-induced changes of forearm blood flow

CONTACTS AND LOCATIONS:
Overall Officials: Walter E Haefeli, MD, Principal Investigator — Heidelberg University
Locations (1):
- DLR Institute of Aerospace Medicine, Cologne, North Rhine-Westphalia, Germany